CLINICAL TRIAL: NCT05995925
Title: Observational Study for Perioperative Care of Patients Requiring ICU (OPICU)
Acronym: OPICU
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Evren Senturk, Prof. Dr., Koç University
Other Study IDs: 2023.198.IRB1.065
Record Dates: First submitted 2023-08-01; First posted 2023-08-16 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Indication, Unlabeled; Complication,Postoperative
Keywords: Intensive Care; Triage; Postoperative period
MeSH Terms: conditions — Postoperative Complications | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with planned ICU admission: Patients with preoperative planned ICU admission
  Interventions: Other: Clinical Observation
- Patients with unplanned ICU admission: Patients with preoperative unplanned ICU admission
  Interventions: Other: Clinical Observation

INTERVENTIONS:
Other: Clinical Observation — Clinical Observation

SUMMARY:
This clinical trial will be carried out as a national multicenter observational cohort trial in Turkey. Our starting point is the need to triage postoperative patients daily due to the limited intensive care unit (ICU) bed capacity. Our hypothesis is that patients requiring emergency or unplanned ICU admission generally meet the ICU admission criteria. However, postoperative patients admitted to the ICU for planned reasons often do not meet the ICU admission criteria and can be monitored in a lower-level unit (Postoperative Care Unit - PACU) for close observation purposes.

The primary aim is to assess the efficient utilization of ICU beds. We try to compare the treatments provided during ICU follow-up, for planned and unplanned patients requiring ICU admission. Our secondary outcome is to identify criteria that can predict ICU indications based on patients' preoperative characteristics and evaluate the postoperative complications according to the Clavien-Dindo classification.

Our aim is to categorize patients admitted to the ICU into two groups: planned and unplanned/emergency cases and compare the necessity of ICU care between these two groups. The need for ICU treatment will be determined based on the criteria established in the following* study. The presence of any of these criteria will indicate the need for ICU admission, while the absence of these criteria may identify patients admitted to the ICU only for monitoring purposes (i.e., unnecessary ICU admissions).

DETAILED DESCRIPTION:
Surgical cases involving patients over 18 years of age requiring postoperative intensive care will be included (including patients who were admitted urgently, or patients that is planned but not admitted to ICU after the surgery).

Cardiac surgery cases, outpatient cases, pediatric surgery cases, patients undergoing surgery while hospitalized in the ICU, patients undergoing only interventional procedures, and those who do not provide consent will be excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Major elective/emergency surgical procedures
* Planned, unplanned, emergent surgical procedures, planned but not admitted to the ICU after the operation.
* Patients who planned but not transferred to the ICU will also be followed/ included postoperatively
* Informed Consent
* Major surgeries will be targeted within the broad subgroup domains of gynecology, neurosurgery, thoracic, urology, orthopedics/trauma, and abdominal surgery.
* Unplanned but admitted to ICU after surgery in 48 hrs.

Exclusion Criteria:

* Day-case surgery
* Cardiac surgery
* Pediatric surgery
* Patients who were already staying in ICU and planned to be operated on
* Denial of informed consent
* All interventional procedures

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients requiring intensive care treatment in the postoperative period.
  The study population comprises individuals who have undergone surgery and require intensive care, regardless of whether their admission to the ICU was planned or unplanned.
Sampling Method: Probability Sample
Enrollment: 1300 (Estimated)
Dates: Start 2024-01-03 (Actual); Primary Completion 2024-02-03 (Estimated); Study Completion 2024-04-03 (Estimated)

PRIMARY OUTCOMES:
Effective use of ICU | From 1 day before the surgery to the 30th day after the surgery.
  To take a picture of the use of ICU beds in postoperative patients in Turkish intensive care units.

SECONDARY OUTCOMES:
Rates of postoperative complications | From the end of the surgery until discharge from the hospital
  They will be assessed postoperatively using Clavien- Dindo classification
Length of ICU stay | From the end of the surgery until discharge from the ICU
  The patient will be followed up from admission to the ICU until discharge from the ICU
Length of hospital stay. | From the end of the surgery until discharge from the hospital
  The patient will be followed up from admission to the ICU until discharge from the hospital
ICU mortality | From the end of the surgery until discharge from the ICU
  The patient will be followed up from admission to the ICU until discharge from the ICU
30-day hospital mortality | From the end of the surgery until discharge from the hospital
  The patient will be followed up from admission to the ICU until his discharge from the hospital
Best scoring system for ICU admission | Preoperative from hospital admission until the patient's discharge from hospital following surgery.
  Identifying the best scoring system for ICU admission by comparing different scoring systems.
Epidemiology of postoperative ICU admitted patients | From preoperative hospital admission until discharge from the hospital
  Defining groups in postoperative patients according to their region or type of surgery
Risk factors or criteria for ICU admission after the surgery | From preoperative hospital admission until discharge from the hospital
  During the entire perioperative process, the patient will be closely observed, vital signs, treatments and complications will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Nahit Cakar, Prof, MD, Study Chair — Koç University
Locations (1):
- Koc University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Result] Jerath A, Laupacis A, Austin PC, Wunsch H, Wijeysundera DN. Intensive care utilization following major noncardiac surgical procedures in Ontario, Canada: a population-based study. Intensive Care Med. 2018 Sep;44(9):1427-1435. doi: 10.1007/s00134-018-5330-6. Epub 2018 Jul 27. PMID 30054691
- [Result] Zampieri FG, Lone NI, Bagshaw SM. Admission to intensive care unit after major surgery. Intensive Care Med. 2023 May;49(5):575-578. doi: 10.1007/s00134-023-07026-7. Epub 2023 Mar 22. No abstract available. PMID 36947198